CLINICAL TRIAL: NCT01426217
Title: Reduction in Intraoperative Lumen Contamination of Standard 3-Way Open Lumen Stopcock Sets Through Use of a Novel, Passive Bundle
Brief Title: Reduction in IV Associated Contamination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: PSI Medical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22743
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Results first posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-08

CONDITIONS: Post-operative Infections
Keywords: IV contamination; intravenous contamination; stopcock contamination; surgical site infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Control arm using standard of care operating room procedures and equipment
- Problem Solving Innovations (PSI) Experimental (Experimental): Implementation of the passive bundle including HubScrub and DocIt
  Interventions: Device: Passive Bundle PSI (Problem Solving Innovations) Medical HubScrub, PSI Medical DocIt

INTERVENTIONS:
Device: Passive Bundle PSI (Problem Solving Innovations) Medical HubScrub, PSI Medical DocIt — Implementation of passive bundle which includes HubScrub and DocIt device into the operating room environment.
  Other Names: PSI Medical HubScrub; PSI Medical DocIt
  Arms: Problem Solving Innovations (PSI) Experimental

SUMMARY:
The purpose of this study is to investigate whether implementing a novel syringe and IV stopcock cap system impregnated with alcohol will reduce IV catheter bacterial contamination and infections in patients.

DETAILED DESCRIPTION:
Bacterial contamination of patient intravenous stopcock sets is a common intraoperative event associated with increased patient mortality, possibly via an infectious mechanism. The most common type of intravenous tubing used in operating rooms is the open lumen stopcock set which lacks a barrier between the environment and intraluminal space, and thus the intravascular space of the patient. The stopcock connector can be easily contaminated by provider hands due to improper handling of the device and/or contaminated by soiled syringe tips subsequently connected to the device. Further, the stopcock connector is often left uncapped by the provider and directly exposed to the environment. Thus, common breaches in intraoperative aseptic practice of healthcare providers can lead to bacterial contamination of the endoluminal space of the open lumen device. The primary aim of the current study is to assess the efficacy of a passive bundle designed to decrease intravenous stopcock and tubing intraluminal bacterial contamination. This passive bundle includes two novel interventions, a DOCit station and HubScrub caps. The HubScrub is designed to clean the needleless connectors and open lumen stopcock systems. The DOCit station is designed to simultaneously clean the interior and exterior of needle-less luer connectors of syringes with isopropyl alcohol while also providing a method of storage and organization of multiple syringes. The investigators hypothesize that the application of this passive bundle to the standard open lumen system commonly employed by anesthesia providers in the operating room will significantly reduce bacterial contamination of standard 3-way open lumen stopcock sets and improve patient safety.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient undergoing surgery or procedure in operating room
* Undergoing general anesthesia

Exclusion Criteria:

* Children (age < 18 years)
* Lack of intravenous access
* failure of anesthesia provider to complete training on experimental device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 594 (Actual)
Dates: Start 2011-08; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan S Brindeiro, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center; Randy W Loftus, MD, Study Director — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Loftus RW, Muffly MK, Brown JR, Beach ML, Koff MD, Corwin HL, Surgenor SD, Kirkland KB, Yeager MP. Hand contamination of anesthesia providers is an important risk factor for intraoperative bacterial transmission. Anesth Analg. 2011 Jan;112(1):98-105. doi: 10.1213/ANE.0b013e3181e7ce18. Epub 2010 Aug 4. PMID 20686007
- [Background] Koff MD, Loftus RW, Burchman CC, Schwartzman JD, Read ME, Henry ES, Beach ML. Reduction in intraoperative bacterial contamination of peripheral intravenous tubing through the use of a novel device. Anesthesiology. 2009 May;110(5):978-85. doi: 10.1097/ALN.0b013e3181a06ec3. PMID 19352154
- [Background] Loftus RW, Koff MD, Burchman CC, Schwartzman JD, Thorum V, Read ME, Wood TA, Beach ML. Transmission of pathogenic bacterial organisms in the anesthesia work area. Anesthesiology. 2008 Sep;109(3):399-407. doi: 10.1097/ALN.0b013e318182c855. PMID 18719437
- [Result] Loftus RW, Brindeiro BS, Kispert DP, Patel HM, Koff MD, Jensen JT, Dodds TM, Yeager MP, Ruoff KL, Gallagher JD, Beach ML, Brown JR. Reduction in intraoperative bacterial contamination of peripheral intravenous tubing through the use of a passive catheter care system. Anesth Analg. 2012 Dec;115(6):1315-23. doi: 10.1213/ANE.0b013e31826d2aa4. Epub 2012 Nov 9. PMID 23144441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted over 3-month period (Aug 1, 2011 to Nov 8, 2011) at Dartmouth-Hitchcock Medical Center, a tertiary care and level 1 trauma center in New Hampshire with 400 inpatient beds and 28 operating suites. The operating rooms enrolled during the study period were randomly selected on a daily basis from the available 28 operating rooms
Groups:
- Experimental Group: Implementation of passive bundle which includes HubScrub and DOCIt device into the operating room environment.
Period: Overall Study
Arm/Group | Control | Experimental Group
Started | 314 | 280
Completed | 306 | 266
Not Completed | 8 | 14
Not completed — lost sample | 8 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental Group | Total
Number analyzed (Participants) | 306 | 266 | 572
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (16.3) | 57.5 (15.7) | 57.6 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 142 | 304
  Male | 144 | 124 | 268
Region of Enrollment [Number; unit: participants]
  United States | 306 | 266 | 572

OUTCOME MEASURES:

1. Primary Outcome: Presence of Bacterial IV Stopcock Lumen Contamination
Description: The presence of bacteria in the stopcock lumen was assessed by analyzing swab cultures of the lumens. Each swab potentially containing bacteria from any of the 3 lumens of the stopcock sets were analyzed
Time Frame: 48 hours
Measure: Number; unit: percent stopcock contamination rate
Units Other Than Participants: Operating Rooms
Groups:
- PSI Experimental: Implementation of passive bundle which includes HubScrub and DocIt device into the operating room environment.
  Problem Solving Innovations (PSI) Passive Bundle: PSI Medical HubScrub, PSI Medical DocIt
Arm/Group | Control | PSI Experimental
Number analyzed (Participants) | 306 | 266
Number analyzed (Operating Rooms) | 306 | 266
percent stopcock contamination rate | 41 | 32
Statistical Analysis 1: Comparison: Control vs PSI Experimental; Test type: Other — Efficacy; Odds Ratio (OR) = 0.79, 95% CI 2-sided [0.63 to 0.98]

2. Secondary Outcome: Presence of Positive Bacterial Culture in IV Stopcock Due to Effluent Contamination
Description: Open lumen ports were removed from the patient; sent directly to the anesthesiology microbiology laboratory; connected by the same clinical laboratory scientist to sterile catheters using sterile, aseptic technique; and injected directly into a BacT/Alert 3D system (bioMérieux Inc., Durham, NC) with 2 mL of sterile saline per port. BacT/Alert is a blood culture system that automatically monitors bacterial growth using colorimetry; a sensor inserted at the bottom of the bottle changes color on detecting the carbon dioxide produced by the growth of the bacteria. Catheters were then removed, and the bottles were directly incubated in the BacT/Alert system for 5 days or until positive. Once positive, the liquid in the bottle was examined to identify the organism.
Time Frame: Until positive, up to 5 days
Population: Specific data for each arm can not be obtained. Sincere efforts were made to obtain and report the data, however, no data is available.
Measure: Number; unit: cases of effluent contamination
Groups:
- Entire Population: Experimental and Control groups were combined for analysis.
  Control arm used standard of care operating room procedures and equipment.
  Experimental arm implemented a of passive bundle which includes HubScrub and DocIt device into the operating room environment.
Arm/Group | Entire Population
Number analyzed (Participants) | 572
cases of effluent contamination | 86
Statistical Analysis 1: Comparison: Entire Population; Test type: Other — Efficacy; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.62 to 1.35]

ADVERSE EVENTS:
Time Frame: 30 days
Description: Experimental & Control groups were combined for analysis. Sincere efforts were made to gather & report data, however, no specific data for each group is available.
  Events:
  * Presence of elevated white blood cells count, fever, anti-infection meds order, office visit/inpatient progress note noting signs of infection &/or bacterial cultures; Positive for ≥1 evaluated if HealthCare Associated Infection
  * Clinical diagnosis of IV catheter-associated phlebitis
Arm/Group | Entire Population
All-Cause Mortality (participants affected / at risk) | 0/572
Serious Adverse Events (participants affected / at risk) | 0/572
Other Adverse Events (participants affected / at risk) | 86/572
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entire Population (N=572)
HCAI (Infections and infestations) | 70 — Healthcare associated infections (HCAI)
Phlebitis (Vascular disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes